CLINICAL TRIAL: NCT06959641
Title: A Phase 2 Open Label Study of XL092 as First Line Therapy in Radioiodine Refractory Differentiated Thyroid Cancer
Brief Title: XL092 for the Treatment of Locally Advanced or Metastatic Radioiodine Refractory Differentiated Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 24N04; NCI-2025-02747 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00223751; NU 24N04 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Locally Advanced Differentiated Thyroid Gland Carcinoma; Locally Advanced Poorly Differentiated Thyroid Gland Carcinoma; Locally Advanced Thyroid Gland Follicular Carcinoma; Locally Advanced Thyroid Gland Oncocytic Carcinoma; Locally Advanced Thyroid Gland Papillary Carcinoma; Metastatic Differentiated Thyroid Gland Carcinoma; Metastatic Poorly Differentiated Thyroid Gland Carcinoma; Metastatic Thyroid Gland Follicular Carcinoma; Metastatic Thyroid Gland Oncocytic Carcinoma; Metastatic Thyroid Gland Papillary Carcinoma; Refractory Differentiated Thyroid Gland Carcinoma; Refractory Poorly Differentiated Thyroid Gland Carcinoma; Refractory Thyroid Gland Follicular Carcinoma; Refractory Thyroid Gland Oncocytic Carcinoma; Refractory Thyroid Gland Papillary Carcinoma; Stage III Differentiated Thyroid Gland Carcinoma AJCC v8; Stage III Thyroid Gland Follicular Carcinoma AJCC v8; Stage III Thyroid Gland Papillary Carcinoma AJCC v8; Stage IV Differentiated Thyroid Gland Carcinoma AJCC v8; Stage IV Thyroid Gland Follicular Carcinoma AJCC v8; Stage IV Thyroid Gland Papillary Carcinoma AJCC v8
MeSH Terms: conditions — Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (XL092) (Experimental): Patients receive XL092 PO QD on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan or MRI and x-ray imaging, and blood and urine sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Survey Administration; Procedure: X-Ray Imaging; Drug: Zanzalintinib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Survey Administration — Ancillary studies
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray
Drug: Zanzalintinib — Given PO
  Other Names: Multi-kinase Inhibitor XL092; XL 092; XL-092; XL092

SUMMARY:
This phase II trial tests how well XL092 works for the treatment of patients with differentiated thyroid cancer that has not responded to previous treatment with radioiodine (radioiodine refractory) and that has spread to nearby tissue or lymph nodes (locally advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). XL092 is in a class of medications called tyrosine kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply, which may help keep cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess efficacy of the treatment zanzalintinib (XL092) in radioiodine refractory/radioactive iodine refractory (RAIR) differentiated thyroid cancer (DTC) patients by evaluating the proportion of patients alive and without progression at 12 months.

SECONDARY OBJECTIVES:

I. Assess efficacy of XL092 treatment in RAIR DTC patients by imaging. II. Assess efficacy of the treatment XL092 in RAIR DTC patients by evaluating progression free survival.

III. Assess efficacy for RAIR DTC patients treated with XL092 evaluating the overall survival time.

IV. Assess the safety and tolerability of XL092 monotherapy in patients with RAIR DTC.

V. Characterize the quality of life in RAIR DTC patients treated with XL092 monotherapy.

EXPLORATORY OBJECTIVES:

I. Assess immune cell landscape in XL092 treated patients. II. Assess by next generation sequencing (NGS) and biomarker analysis, mechanisms that lead to response or failure to XL092.

OUTLINE:

Patients receive XL092 orally (PO) daily (QD) on days 1-21 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) and x-ray imaging, and blood and urine sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days then every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed locally advanced or metastatic, radioactive iodine (RAI) refractory, differentiated thyroid cancer (including papillary, follicular, and oncocytic/Hurthle cell, and poorly differentiated thyroid cancer [PDTC]), with progression within 12 months (per Response Evaluation Criteria in Solid Tumors [RECIST] version [v] 1.1 response criteria) prior to study registration, and no prior therapy in the RAI-refractory setting and for which standard curative or palliative measures do not exist or are no longer effective.

  * NOTE: RAI refractoriness is defined as absence of uptake of RAI on either a low-dose diagnostic test or a post-treatment RAI scan in measurable lesions or radiographic progression of disease within 12 months of the last course of RAI treatment despite the recorded uptake of RAI with that previous therapy or having a cumulative lifetime administered dose of ≥ 600mCi.
  * Poorly differentiated thyroid cancer (PDTC) is typically classified as a type of differentiated thyroid cancer (as opposed to undifferentiated thyroid cancer or anaplastic thyroid cancer)
* Patients must have measurable disease according to RECIST v 1.1
* Patients must be age ≥ 18 years
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2
* Leukocytes (WBC) ≥ 3,000/mcL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL

  * Prophylactic use of granulocyte colony-stimulating factor (G-CSF) will not be allowed within 2 weeks of relevant screening laboratory testing. However, G-CSF may be employed in accordance with current American Society of Clinical Oncology (ASCO) guidelines for treatment-emergent neutropenia observed at any time during the study
* Hemoglobin (Hgb) ≥ 9 g/dL

  * Prophylactic use of blood transfusions for anemia and thrombocytopenia is not allowed within 2 weeks prior to relevant screening laboratory testing, but such treatment is allowed for treatment-emergent anemia or thrombocytopenia, as indicated by the current ASCO and American Association of Blood Banks guidelines
* Platelets (PLT) ≥ 100,000/mcL

  * Prophylactic use of blood transfusions for anemia and thrombocytopenia is not allowed within 2 weeks prior to relevant screening laboratory testing, but such treatment is allowed for treatment-emergent anemia or thrombocytopenia, as indicated by the current ASCO and American Association of Blood Banks guidelines
* Total bilirubin ≤ 1.5 x Institutional upper limit of normal (ULN) ; for subjects with Gilbert's disease ≤ 3 x ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 3 x Institutional ULN
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x Institutional ULN
* ALP (alkaline phosphatase) ≤ 3 x Institutional ULN; For subjects with documented bone metastasis, ≤ 5 x ULN
* Creatinine Clearance (CrCl) ≥ 40 mL/min (≥ 0.67 mL/sec) using the Cockcroft-Gault equation
* International Normalized Ratio (INR) ≤ 1.5 x Institutional ULN (in patients not currently on therapeutic anticoagulation)
* Activated partial thromboplastin time (aPTT) ≤ 1.2 × Institutional ULN (in patients not currently on therapeutic anticoagulation)
* Urine protein-to creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.1 mg/mmol)
* For patients with a known history of human immunodeficiency virus (HIV), infected patients on effective anti-retroviral therapy must have a viral load undetectable for 6 months prior to registration. Please note this lab is not a requirement for eligibility, however, if it has been completed previously as part of the patient's health care, it should be documented for eligibility.

  * NOTE. To be eligible, patients must not have known uncontrolled infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
  * NOTE: patients must meet all of the following criteria:

    * On stable anti-retroviral therapy
    * CD4+ T cell count ≥ 200/µL; and
    * An undetectable viral load.
  * NOTE: HIV testing will be performed at screening if it is required by local regulation or per standard of care (SOC).
  * NOTE: To be eligible, patients taking CYP inhibitors (e.g., zidovudine, ritonavir, cobicistat, didanosine) or CYP3 inducers (efavirenz) must change to a different regimen not including these drugs 7 days prior to initiation of study treatment. Anti-retroviral therapies (ART) must have been received for at least 4 weeks prior to the first dose.
  * NOTE: CD4+ T cell counts, and viral load are monitored per standard of care by the local health care provider
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and patients are stable for at least 4 weeks before the first dose of study treatment.

  * NOTE: Patients with active brain metastases are not allowed.
  * NOTE: Therapeutic doses of Low Molecular Weight Heparin (LMWH) are not permitted in patients with known brain metastases
* Patients of child-bearing potential must have a negative pregnancy test prior to registration on study.

  * NOTE: Patients of child-bearing potential are considered to be of child-bearing potential unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 consecutive months of amenorrhea in a patient of child-bearing potential > 45 years-of-age in the absence of other biological or physiological causes). In addition, a patient of child-bearing potential < 55 years-of-age must have a serum follicle stimulating hormone (FSH) level > 40 mIU/mL to confirm menopause)
* The effects of XL092 on the developing human fetus are unknown. For this reason and because tyrosine kinase inhibitors (TKIs) as well as other therapeutic agents used in this trial are known to be teratogenic, sexually active fertile patients and their partners must agree to use highly effective methods of contraception during the course of the study and for the following durations after the last dose of study treatment (whichever is later): Through 186 days after the last dose of XL092 for patients of child-bearing potential or through 96 days after the last dose of XL092 for patients of sperm producing capacity. Because the effect of XL092 on the pharmacokinetics (PK) of contraceptive steroids has not been investigated, hormonal contraceptives may not achieve the level considered "highly effective". For this reason, an additional contraceptive method, such as a barrier method (e.g., condom), may be required. In addition, patients of sperm producing capacity must agree not to donate sperm and patients of child-bearing potential must agree not to donate eggs (ova, oocyte) for the purpose of reproduction during these same periods. Should a patient of child-bearing potential become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately
* Recovery to baseline or ≤ grade 1 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5 from adverse events (AE[s]) related to any prior treatments unless AE(s) are deemed clinically nonsignificant by the Treating Investigator and/or stable on supportive therapy.

  * NOTE: Patients must have recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) except for alopecia, neuropathy, and other non-significant adverse events per NCI CTCAE v 5.0
* Patients must have the ability to understand and the willingness to sign a written informed consent document and comply with the protocol requirements
* Patients must have the ability to swallow, retain and absorb oral medications

  * NOTE: Patients must have the ability to swallow tablets or ingest a suspension either orally or by a nasogastric (NG) or gastrostomy (PEG) tube

Exclusion Criteria:

* Prior treatment with XL092 (zanzalintinib)
* Patient has hepatitis B
* Patient has hepatitis C.

  * NOTE: Patients with treated hepatitis C and positive hepatitis C virus (HCV) antibody test are eligible only if followed by a negative HCV ribonucleic acid (RNA) test and no ongoing anti-HCV therapy. The HCV RNA test will be performed only for patients who have a positive HCV antibody test
* Patient is pregnant or nursing (lactating)

  * NOTE: Pregnant patients are excluded from this study because XL092 is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with XL092, breastfeeding should be discontinued if the mother is treated with XL092
* Receipt of any type of small molecule kinase inhibitor treatment (including investigational kinase inhibitor) within 2 weeks before the first dose of study treatment
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational therapy or investigational device) within 4 weeks before the first dose of study treatment.

  * NOTE: For patients that received nitrosoureas or mitomycin C, < 6 weeks prior to planned treatment start date
* Radiation therapy for bone metastases within 2 weeks, any other radiation therapy within 4 weeks before the first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment.

  * NOTE: Patients with clinically relevant ongoing complications from prior radiation therapy are not eligible
* Previously identified allergy or hypersensitivity to components of the study treatment formulations, have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to XL092 (zanzalintinib)
* Concomitant anticoagulation with oral anticoagulants (e.g., warfarin or other coumarin-related agents, direct thrombin inhibitors, or anti-platelet agents such as clopidogrel, chronic use of aspirin above low dose levels for cardio-protection per institutional practice).

  * NOTE: Allowed anticoagulants are the following: prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low molecular weight heparins (LMWH); Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.
  * NOTE: Patients must have discontinued oral anticoagulants within 3 days or 5 half-lives prior to first dose of study treatment, whichever is longer.
  * NOTE: Therapeutic doses of LMWH are not permitted in subjects with known brain metastases
* Any complementary medications (e.g., herbal supplements or traditional Chinese medicines) to treat cancer within 2 weeks before first dose of study treatment
* Patient has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 3 or 4, Class 2 or higher, unstable angina pectoris, new-onset angina, serious cardiac arrhythmias (e.g., ventricular flutter, ventricular fibrillation, Torsades de pointes).
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant ischemic event within 6 months before first dose of study treatment.
    * Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous or non-cerebrovascular accident (CVA)/TIA arterial thromboembolic events within 3 months before the first dose of study treatment.

      * NOTE: Patients with a diagnosis of DVT within 6 months are allowed if asymptomatic and stable at screening and treated with anticoagulation per standard of care for at least 1 week before the first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen.
      * NOTE: Patients who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator.
    * Prior history of myocarditis
  * Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

    * Tumors invading the GI-tract from external viscera
    * Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis
    * Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months unless cause of obstruction is definitively managed and patient is asymptomatic
    * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose.

      * NOTE: Complete healing of an intra-abdominal abscess must be confirmed before the first dose of study treatment.
    * Known gastric or esophageal varices
    * Ascites, pleural effusion, or pericardial fluid requiring drainage in the last 4 weeks
* Other clinically significant disorders that would preclude safe study participation including having an uncontrolled intercurrent illness including, but not limited to any of the following:

  * Ongoing or active infection requiring systemic treatment

    * NOTE: Prophylactic antibiotic treatment is allowed (e.g. for uncomplicated infections such as urinary tract infections [UTIs] or sinus infections being treated with oral antibiotics)
  * Serious non-healing wound/ulcer/bone fracture.

    * NOTE: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions
  * Patient has malabsorption syndrome
  * Pharmacologically uncompensated, symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ or allogeneic stem cell transplant.
  * Any other illness or condition or laboratory finding that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment
* Symptomatic cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.

  * NOTE: Asymptomatic or radiated endobronchial disease lesions allowed
* Lesions invading major blood vessel(s), including, but not limited to, inferior vena cava, pulmonary artery, or aorta

  * NOTE: Subjects with intravascular tumor extension (e.g., tumor thrombus in renal vein or inferior vena [V.] cava) may be eligible following Principal Investigator approval
* Major surgery e.g., GI surgery, removal, or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Prior laparoscopic surgeries (i.e., nephrectomy) within 4 weeks prior to first dose of study treatment. Minor surgery (e.g., simple excision, tooth extraction) within 5 days before the first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to the first dose of study treatment.

  * NOTE: Fresh tumor biopsies should be performed at least 5 days before the first dose of study treatment for screening procedures.
  * NOTE: Patients with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms within 14 days per electrocardiogram (ECG) before first dose of study treatment.

  * NOTE: electrocardiogram (ECG) evaluation is required at screening; QT prolongation is a potential side effect of VEGFR-associated TKIs, such as XL092
* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent
* Patients with:

  * Any other active malignancy within 2 years prior to start of study treatment
  * A prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
  * NOTE: Allowed: Superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy. Incidentally diagnosed prostate cancer is allowed if assessed as stage ≤ T2N0M0 and Gleason score ≤ 6
* Administration of a live, attenuated vaccine (e.g., Intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin, yellow fever, varicella, and TY21a typhoid vaccines) is prohibited:

  * Within 30 days before the first dose of study treatment and
  * Prohibited for all patients while on study treatment

    * NOTE: Experimental vaccines are not allowed while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-09-11 (Estimated); Study Completion 2030-09-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the time of the first dose of XL092 to the first documentation of disease progression, initiation of subsequent anti-cancer therapy, completion of 12 months of participation, or death from any cause, whichever occurs first, assessed at 12 months
  Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria. Median PFS at 12-months will be analyzed using the Kaplan-Meier method. The 12-month PFS estimate will be reported along with the confidence interval. Cox proportional hazards models will be applied to assess the impact of covariates such as age, sex, baseline disease severity, and genetic markers on PFS, when appropriate.

SECONDARY OUTCOMES:
Radiographic response rate | Up to 12 month follow-up
  Defined as the proportion of patients who achieve a complete response or partial response as per RECIST v1.1. The point estimate of the objective response rate will be reported with its 2-sided 95% Clopper-Pearson exact confidence interval.
Overall PFS | From the first dose of XL092 to the date of the first progression event or death from any cause, assessed up to 12 month follow-up
  Will use the Kaplan-Meier method to estimate the overall PFS distribution. Subgroup comparisons will be made using log-rank tests, and a Cox proportional hazards model will be employed to assess covariate effects.
Overall survival (OS) | From the start of treatment with XL092 to the date of death from any cause, assessed up to 12 month follow-up
  OS will also be analyzed using the Kaplan-Meier estimator. Differences in survival distributions across patient subgroups will be evaluated using log-rank tests, and Cox models will be used to explore the effects of demographic and clinical variables on OS.
Incidence of adverse events | Up to 30 days after the end of treatment
  Assessed by clinical review of all relevant parameters, including adverse events (AEs), concomitant medication queries, Eastern Cooperative Oncology Group performance status, weight and vital signs measurements, electrocardiogram measurements, and clinical laboratory testing values. The severity of AEs will be graded as mild, moderate, severe, or life-threatening according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. All reported toxicities, regardless of attribution, by toxicity type and maximum grade will be summarized, and sorted by number of patients experiencing the toxicity. The maximum grade consolidates the reports of a given toxicity for a patient over time by taking the maximum across time. Categorical data analyses and summary statistics will be used to report AEs.
Changes in quality of life | Baseline to 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jochen H Lorch, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States